CLINICAL TRIAL: NCT04861896
Title: An e-Health Intervention to Improve Symptom Burden and Health-Related Quality of Life Among Hispanic Women Completing Active Treatment for Breast Cancer
Brief Title: A Research Study for Latina Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Betina Yanez, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00201961B
Record Dates: First submitted 2021-03-31; First posted 2021-04-27 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Cancer, Breast; Cancer-related Problem/Condition; Quality of Life; Hormone Dependent Neoplasms; Adherence, Medication
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Hormone-Dependent; Medication Adherence | interventions — Self-Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "My Guide" (psychoeducation & self management program) (Experimental): Smartphone-based program plus standard clinical care.
  Interventions: Behavioral: "My Guide" (psychoeducation & self-management program)

INTERVENTIONS:
Behavioral: "My Guide" (psychoeducation & self-management program) — 12-week long health promotion Smartphone application to support patient's side effects self-management and adherence to endocrine therapy.

SUMMARY:
The purpose of this study is to examine the feasibility and preliminary efficacy of a psychosocial eHealth intervention designed to improve hormone therapy adherence among Hispanic/Latinx women with breast cancer. Our proposed secondary outcomes are health-related quality of life and self-efficacy in managing hormone therapy side effects.

The intervention components include breast cancer knowledge, hormone/endocrine therapy knowledge, stress awareness and management, social support, and enhanced communication and intimacy skills. The intervention will be delivered via a Smartphone application over a 12-week period.

All participants will receive the intervention application (described below). Aside from using the Smartphone application for the recommended 12 weeks, participation in this study includes three assessments: baseline (at the beginning of the research study), 6-week follow-up, and 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of breast cancer, non-metastatic, stage 0-III (A, B, or C)
* Receiving or received endocrine/hormone therapy within the last 3 years (36 months)
* At least 18 years of age
* Able to speak and read English or Spanish
* Able to provide informed consent
* Self-identify Hispanic/Latina ethnicity

Exclusion Criteria:

* Stage IV or metastatic
* Visual, hearing, voice, or motor impairment that would prevent completion of study procedures
* Diagnosis of an unmanaged psychotic disorder, bipolar disorder, dissociative disorder, or other diagnoses for which participation in this trial is either inappropriate or dangerous - this includes patients who have a life-threatening illness (e.g., end-stage kidney disease) or diagnosis of a chronic disease that is associated with a major functional impairment (e.g., fibromyalgia)
* Illicit substance or alcohol dependence
* Suicidal ideation, plan, intent
* Alzheimer's, dementia, or history of stroke
* Scheduled reconstruction surgery within 1 month of any study procedures or involvement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Acceptability of My Guide: Usefulness | T3 (immediately following 12 week intervention)
  To assess acceptability, all participants are asked to complete an exit interview on My Guide. This interview assesses usefulness, satisfaction, learnability and usability of the application. This exit interview was synthesized from validated measures assessing eHealth intervention acceptability, and was adapted for our study to better fit our target population and our application design. Above average scores on the questionnaire are considered acceptable. The questionnaire is administered over the phone immediately following the 12 week intervention.
Acceptability of My Guide: Satisfaction | T3 (immediately following 12 week intervention)
  To assess acceptability, all participants are asked to complete an exit interview on My Guide. This interview assesses usefulness, satisfaction, learnability and usability of the application. This exit interview was synthesized from validated measures assessing eHealth intervention acceptability, and was adapted for our study to better fit our target population and our application design. Above average scores on the questionnaire are considered acceptable. The questionnaire is administered over the phone immediately following the 12 week intervention.
Acceptability of My Guide: Learnability | T3 (immediately following 12 week intervention)
  To assess acceptability, all participants are asked to complete an exit interview on My Guide. This interview assesses usefulness, satisfaction, learnability and usability of the application. This exit interview was synthesized from validated measures assessing eHealth intervention acceptability, and was adapted for our study to better fit our target population and our application design. Above average scores on the questionnaire are considered acceptable. The questionnaire is administered over the phone immediately following the 12 week intervention.
Acceptability of My Guide: Usability | T3 (immediately following 12 week intervention)
  To assess acceptability, all participants are asked to complete an exit interview on My Guide. This interview assesses usefulness, satisfaction, learnability and usability of the application. This exit interview was synthesized from validated measures assessing eHealth intervention acceptability, and was adapted for our study to better fit our target population and our application design. Above average scores on the questionnaire are considered acceptable. The questionnaire is administered over the phone immediately following the 12 week intervention.
Demand of My Guide: Recruitment Rate | 12 weeks
  We assess demand of the My Guide application through study recruitment. Based on previous psychosocial and behavioral studies in oncology, an 70% recruitment rate is considered an adequate level of demand.
Demand of My Guide: Retention Rate | 12 weeks
  Another way we assess demand of the My Guide application is through participant retention. Based on previous psychosocial and behavioral studies in oncology, an 70% retention rate is considered an adequate level of demand.
Participant use of My Guide: Number of Login's | 12 weeks
  We assess participant use of the My Guide application by examining the number of participant logins to the web-based application.
Participant use of My Guide: Duration of Usage | 12 weeks
  We assess participant use of the My Guide application by examining the duration participant time spent on the website. Based on previous psychosocial and behavioral studies in oncology, an average of 8 hours of use is considered an adequate level of engagement.
Participant use of My Guide: Content Accessed | 12 weeks
  We assess participant use of the My Guide application by examining the type of content accessed by participants on the website.
Change in Medication adherence will be assessed primarily with the Adherence to Refills and Medication Scale (ARMS). | T1 (prior to starting intervention), T2 (6 weeks into intervention), T3 (immediately following 12 week intervention)
  The ARMS (Adherence to Refills and Medications Scale) survey is a previously validated patient-report measure of barriers to medication adherence and adherence-related behavior.

SECONDARY OUTCOMES:
Change in Health Related Quality of Life will be evaluated with The Functional Assessment of Cancer Therapy (FACT-G7) | T1 (prior to starting intervention), T2 (6 weeks into intervention), T3 (immediately following 12 week intervention)
  The FACT-G7 is a validated questionnaire that assesses top-rated symptoms and concerns for a broad spectrum of advanced cancers and serves as a health-related quality of life (HRQoL) measure.
Change in Patient Self-Efficacy in managing side effects is measured using the PROMIS Self Efficacy for Managing Symptoms | T1 (prior to starting intervention), T2 (6 weeks into intervention), T3 (immediately following 12 week intervention)
  The PROMIS Self Efficacy for Managing Symptoms survey is a validated, computer adaptive survey to assess how confident participants are in their ability to manage their symptoms and side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States